CLINICAL TRIAL: NCT04629924
Title: Comparison of Intraosseous Anesthesia Osteocentral With Electronic Assistance to Injection to a Conventional Anaesthesia by Infiltration on Temporary Molars
Brief Title: Comparison of Intraosseous Anesthesia Osteocentral With Electronic Assistance to Injection With Conventional Anesthesia
Acronym: SLEEPER-ONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20-AOI-06
Record Dates: First submitted 2020-11-10; First posted 2020-11-16 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2022-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This is a multicentre, randomized, split-mouth, randomized controlled trial in which the experimental and control anesthetic systems will be randomly assigned to the teeth (randomization unit) of the tooth pair. controlerals considered in the same patient. This design allows a gain in power, each subject being its own witness without any carry-across effect, the two treatments being separated by one to two weeks ("split-mouth cross-over").
Who Masked: Participant, Outcomes Assessor
Masking Description: The dental surgeon cannot, of course, be blind to the type of anesthesia. The subject may be kept blind to the type of anesthesia administered. This is the most important since the main criterion of judgment is a criterion reported by the patient (his or her pain during anesthesia). Similarly, the evaluator will be kept blind to the type of anesthesia administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sleeper one (Experimental): Topical anesthesia: to be applied during 1 to 2 minutes on a previously dried mucous membrane (Lidocaine Gingival Gel, Septodont).
  Osteocentral anesthesia performed with the SleeperOne® 5 system (Dental Hi Tec) loaded with Articaine 1/200000 carpule.
  Interventions: Device: sleeper one; Device: conventional technis
- conventional technique (Active Comparator): Topical anesthesia: to be applied during 1 to 2 minutes on a previously dried mucous membrane (Lidocaine Gingival Gel, Septodont).
  Anaesthesia using a conventional technique, i.e. a metal syringe loaded with Articaine 1/200000 carpule.
  Interventions: Device: sleeper one; Device: conventional technis

INTERVENTIONS:
Device: sleeper one — anesthesic injection with sleeper one device
Device: conventional technis — anesthesic injection with the conventional technic

SUMMARY:
Anesthesia systems with electronic injection assistance for slow injection pressure-limiting drips (especially for intraosseous anaesthesia) are offered to limit pain. The European Academy of Pediatric Dentistry (EAPD) recommends them for their pen-like appearance which avoids the negative aspect of the classic syringe (Kühnisch 2017). A review systematic review of the literature (Smolarek et al 2019) including 20 randomized controlled trials conducted at children and adolescents showed a significant reduction in pain with the systems with electronic assistance compared to conventional anaesthesia performed with a syringe (-0.8: IC95% (-1.3, -0.3)). Only four of them (Tahmassebi et al 2009, Kandiah and Tahmassebi 2012, Patini et al 2018, Smail-Faugeron et al 2019) were at low risk of bias, and only two parallel group trials were of poor quality and included only children in temporary dentition in which anaesthesia, often problematic, was performed only in the maxilla (Allen et al 2002, Klein et al, 2005) without assessing the intensity of the pain felt.

(FPS-R).

The tested strategy, anesthesia system with electronic injection assistance (SleeperOne® 5 Dental Hi Tec), compared to a conventional metallic anaesthetic syringe currently considered as the standard for performing local anesthesia during oral treatments painful, meets the ISO 13485: 2016 standard.

Elements justifying that the particular surveillance modalities added by research do not involve negligible risks and constraints

Specific monitoring modalities added by research include :

* Explanation of the study to each eligible child and his or her legal guardians
* Gathering the informed consent of the child and his or her legal guardians
* The determination of comparative anesthesia systems (SleeperOne® 5 versus syringe metal)
* Data collection during the two care sessions (maximum 15 days apart)

It is a use of a product placed on the market whose conditions of use are in conformity with its destination and its current conditions of use (RIPH Category 2 application decree) There is no additional consultation or visit, nor any additional examination, in relation to the management in accordance with the recommendations of good practice of a child affected by a carious disease corresponding to the children included. On the other hand, the consultation will take a little longer due to the indicators to be collected and the data entry. These particular surveillance modalities added by research have only negligible constraints.

ELIGIBILITY:
Inclusion Criteria:

* Written consent of one of the two parents (legal guardians) and the child,
* Child and parents (legal guardians) speaking French,
* Child covered by his parents' social security coverage,
* Child aged 4-8 years in temporary stable denture,
* Child in good general health (ASAI or II),
* Child cooperating in care in the vigilant state (cooperation evaluated with a Venham score) 0, 1, 2).
* Child with two temporary molars of the same type, 1st or 2nd molars, controlateral (fractional mouth test) belonging to different quadrants of the the same arch (pair of teeth 54-64, 55-65, 74-84 or 75-85) and each requiring a single equivalent conservative treatment under anaesthesia (ICDAS 3 to 6 carious lesions on teeth) vital).

Exclusion Criteria:

They are declined at the scale of the subject and the tooth:

* Child having taken an analgesic treatment 24 hours before randomization,
* Child allergic to local anesthetics
* Child with at least one of the two temporary molars of the same pair (54-64, 55-65, 74-84 or 75-85) has inflammatory or infectious complications (symptomatology of irreversible pulpitis, clear radio image) and in front of this fact to make the object of a pulpectomy or avulsion :
* Molar presenting spontaneous pain outside of meals or continuous pain.
* Temporary molar whose radiographic examination reveals an enlargement of the space desmodontal, the presence of a radio-clear image at the furcation and/or the periapical regions, or even internal or external resorption.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-11-24 (Actual)

PRIMARY OUTCOMES:
patient pain | 18 months
  intensity of pain felt by the patient according to the face scale.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Lille University Hospital, Lille
  - Nantes University Hospital, Nantes
  - Nice Hospital, Nice
  - Rennes University Hospital, Rennes
  - Toulouse university Hospital, Toulouse